CLINICAL TRIAL: NCT03891576
Title: A Multicenter, Open-label Phase II Trial of a New Customized Dosing (RADAR Dosing) of Niraparib As Maintenance Therapy in Platinum Sensitive Ovarian, Fallopian Tube or Primary Peritoneal Recurrent Cancer Patients
Brief Title: Newton Study (NEW Dosing MainTenance Therapy Ovarian CaNcer)
Acronym: Newton
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: North Eastern German Society of Gynaecological Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRFMN-OVA-7814
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; Platinum Senitive; Recurrent Cancer; Niraparib; Thrombocytopenia; Neutropenia; Anemia; RADAR dosing; Maintenance Therapy; PARP-inhibitor
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Recurrence; Thrombocytopenia; Neutropenia; Anemia | interventions — niraparib

STUDY DESIGN:
Intervention Model Description: This is a study built up by a randomized and a no-randomized part.
  Randomized part:
  Patients who either have a baseline body weight ≥58 and <77kg, or have a baseline body weight ≥77kg and baseline platelet count <150,000/µL (named as restricted population) will be randomly assigned to receive RADAR dosing or the SmPC dosing.
  Randomization ratio will be 1:1 and will be based on a minimization procedure accounting for the following factors: i. platinum sensitivity; ii. use of bevacizumab in conjunction with the penultimate platinum based therapy; iii. best response (complete or partial) during the last platinum regimen.
  No-randomized part:
  Patients with weight <58 or ≥77kg and baseline platelet count ≥150,000/µL will be enrolled into the study but not randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Niraparib 200 mg (Experimental): Niraparib will be administered every day as oral at a fixed dose of 200 mg
  Interventions: Drug: Niraparib
- Niraparib 300 mg (Active Comparator): Niraparib will be administered every day as oral at a fixed dose of 300 mg
  Interventions: Drug: Niraparib
- Niraparib 200mg/300mg (Other): Niraparib will be administered every day as oral at a fixed dose of 200 mg or 300 mg
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib is a potent, orally active PARP1 and PARP2 inhibitor being developed as a treatment for patients with tumors that harbor defects in the homologous recombination DNA repair pathway or that are driven by PARP-mediated transcription factors.
  Other Names: Zejula

SUMMARY:
This study evaluates whether the adoption of the RADAR dosing strategy could further reduce treatment related toxicities improving the safety profile of niraparib.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older, female, any race
2. Histologically diagnosed ovarian cancer, fallopian tube cancer or primary peritoneal cancer
3. High grade (or grade 3) serous histology or known to have gBRCAmut
4. Has received at least 2 previous lines of platinum-containing therapy (not necessarily consecutive), and has disease that was considered platinum sensitive following the penultimate platinum line (more than 6-months period between penultimate platinum regimen and progression of disease)
5. Has responded to the last platinum line (PR or CR)
6. No more than 8 weeks have elapsed from completion of the last platinum regimen and the patient is still not progressing after response
7. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
8. Adequate bone marrow, kidney and liver function, defined as follows:

   1. Absolute neutrophil count ≥ 1,500/µL
   2. Platelets ≥ 100,000/µL
   3. Hemoglobin ≥ 9 g/dL
   4. Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault equation
   5. Total bilirubin ≤ 1.5 x ULN (≤2.0 in patients with known Gilberts syndrome) OR direct bilirubin ≤ 1 x ULN
   6. Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN unless liver metastases are present, in which case they must be ≤ 5 x ULN
9. Patient receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy.
10. Patient must have a negative urine or serum pregnancy test within 7 days prior to taking study treatment if childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment or use adequate barrier methods throughout the study. Non-childbearing potential is defined as follows (by other than medical reasons): ≥45 years of age and has not had menses for >1 year; patients with amenorrhea for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation; Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 180 days after the last dose of study treatment.
11. Patient must agree to not breastfeed during the study or for 180 days after the last dose of study treatment.
12. Patient must be able to understand the study procedures and agree to participate in the study by providing written informed consent.
13. Patients must have normal blood pressure or adequately treated and controlled hypertension. (i.e. systolic BP ≤ 140 mmHg and diastolic BP ≤ 90 mmHg)

Exclusion Criteria:

1. Patient simultaneously enrolled in any interventional clinical trial
2. Invasive cancer other than ovarian cancer within 2 years (except basal or squamous cell carcinoma of the skin that has been definitely treated)
3. Patient with known, symptomatic brain or leptomeningeal metastases
4. Patient with immunocompromised status
5. Patient with known active hepatic disease
6. Prior treatment with a known PARP inhibitor
7. Patient who has had major surgery ≤ 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects.
8. Patient who has received investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy.
9. Patient has had radiation therapy encompassing >20% of the bone marrow within 2 weeks prior to day 1 of protocol therapy
10. Patient has had any radiation therapy within 1 week prior to day 1 of protocol therapy.
11. Patient with known hypersensitivity to niraparib components or excipients.
12. Patient has received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy.
13. Patient has received colony stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy.
14. Patient has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
15. Patient with any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
16. Patient with a serious, uncontrolled medical disorder. Examples include, but are not limited to, nonmalignant systemic disease, active, uncontrolled infection, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Safety: Occurrence of grade ≥3 thrombocytopenia | 3 months
  Rate of patients experiencing a grade ≥3 thrombocytopenia during the first three cycles

SECONDARY OUTCOMES:
Safety: Occurrence of grade ≥ 3 thrombocytopenia | 6 months
  Rate of patients experiencing a grade ≥3 thrombocytopenia during the first six cycles
Safety: Maximum toxicity grade | Up to two years after the last patient enrolled
  Maximum toxicity grade experienced by each patient, for each toxicity, according to NCI-CTCAE v. 4.03
Safety: Grade 3-4 toxicities | Up to two years after the last patient enrolled
  Patient experiencing grade 3-4 for each toxicity
Safety: SAE | Up to two years after the last patient enrolled
  Type, frequency and nature of SAEs
Safety: Number of patients with at least a SAE | Up to two years after the last patient enrolled
  Number of patients with at least a SAE
Safety: Number of patients with at least a SADR | Up two years after last patient enrolled
  Number of patients with at least a SADR
Safety: Number of patients with at least a SUSAR | Up two years after last patient enrolled
  Number of patients with at least a SUSAR
Efficacy: PFS-6 | 6 months
  PFS rate at 6 months, defines as the proportion of patients alive and free from progression at 6 months after randomization
Efficacy: PFS | Up two years after last patient enrolled
  PFS, defined as the time from the date of treatment randomization to the date of first documentation of progression or death whichever occurs first
Efficacy: OS | Up two years after last patient enrolled
  OS at 24 months, defined as the rate of patients who are alive at 24 months from randomization
Pharmacokinetic | Up to two years after the last patient enrolled
  Trough level of niraparib concentration at steady state (Css) and peak level at 2 hours after dosing
Compliance | Up to two years after the last patient enrolled
  Number of administered cycles
Compliance | Up to two years after the last patient enrolled
  Frequency and reasons for drug discontinuation and treatment modification
Compliance | Up to two years after the last patient enrolled
  Dose intensity

CONTACTS AND LOCATIONS:
Overall Officials: Nicoletta Colombo, MD, Principal Investigator — Istituto Europeo di Oncologia (IEO) - Milan
Locations (12):
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - University Hospital Dresden, Dresden
  - Kliniken Essen Mitte, Essen
- Italy (9):
  - ASST degli Spedali Civili di Brescia, Brescia
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale dei Tumori, Milan
  - Ospedale San Gerardo, Monza
  - Istituto Oncologico Veneto (IOV), Padua
  - AO Arcispedale Santa Maria Nuova, Reggio Emilia
  - Policlinico Umberto I, Università di Roma "La Sapienza", Roma
  - AO Ordine Mauriziano, Torino
  - AOU Città della Salute e della Scienza di Torino - Ospedale Sant'Anna, Torino

IPD SHARING:
Plan to Share IPD: No